CLINICAL TRIAL: NCT05163353
Title: Prospective, Multicenter, Controlled, Evaluator-blind, Randomized Study to Investigate the Effectiveness and Safety of Diluted RADIESSE® for Treatment of Décolleté Wrinkles
Brief Title: Evaluation of the Effectiveness and Safety of Diluted RADIESSE® in the Treatment of Décolleté Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M930521003
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Décolleté Wrinkles
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment with diluted Radiesse (Experimental): Injection of Décolleté Wrinkles with diluted Radiesse
  Interventions: Device: Treatment with diluted Radiesse
- Delayed treatment with diluted Radiesse (Other): Delayed injection of Décolleté Wrinkles with diluted Radiesse
  Interventions: Device: Treatment with diluted Radiesse

INTERVENTIONS:
Device: Treatment with diluted Radiesse — Injection of Décolleté Wrinkles with diluted Radiesse

SUMMARY:
Trial to confirm the effectiveness and demonstrate the safety of treatment with diluted Radiesse for correction of Décolleté Wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* Female between ≥ 30 and ≤ 65 years old at the time of the screening.
* Subjects seeking improvement of décolleté wrinkles.

Exclusion Criteria:

* Any previous surgery, including plastic surgery or permanent surgical implant in the treatment area.
* Previous treatment with collagen fillers, calcium hydroxylapatite, and/or long-lasting hyaluronic acid (HA) fillers in the décolleté, or with other HA fillers in the décolleté.
* Previous treatment with botulinum toxin, ablative or fractional laser, microdermabrasion, microneedling, chemical peels, and/or non-invasive skin tightening in the décolleté.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2025-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Clinical Testing of Beverly Hills, Merz Investigational Site #0010395, Beverly Hills, California
  - Facial Plastic Surgery, Merz Investigational Site #0010463, Redondo Beach, California
  - Cosmetic Laser Dermatology, Merz Investigational Site #0010321, San Diego, California
  - Private Practice, Merz Investigational Site #0010299, Santa Monica, California
  - Face Beautiful Inc, Merz Investigational Site #0010358, Vista, California
  - Skin Associates of South Florida, Merz Investigational Site #0010101, Coral Gables, Florida
  - Research Institute of the Southeast, LLC, Merz Investigational Site #0010420, West Palm Beach, Florida
  - The Graivier Center, Merz Investigational Site #0010464, Alpharetta, Georgia
  - Nashville Center for Laser and Facial Surgery, Merz Investigational Site #0010353, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 9 investigational sites in the United States.
Pre-assignment Details: A total of 152 subjects were enrolled and randomized in the study.
Groups:
- Treatment With Radiesse: Subjects received three injections of diluted Radiesse using cannula in the décolleté treatment area on Day 1, Week 6, and Week 12. Subjects were eligible to receive an optional retreatment at Week 36.
- Untreated Control/Delayed Treatment With Radiesse: Subjects remained untreated until Week 24 and then received three injections of diluted Radiesse using cannula in the décolleté treatment area at Week 24, Week 30, and Week 36. Subjects in this group had no option of retreatment.
Period: Overall Study
Arm/Group | Treatment With Radiesse | Untreated Control/Delayed Treatment With Radiesse
Started | 116 | 36
Intent to Treat (ITT) Set (ITT population included all randomized subjects.) | 116 | 36
Safety Evaluation Set (SES) (9 subjects randomized in "Treatment With Radiesse" group and 6 subjects randomized in "Untreated Control/Delayed Treatment With Radiesse" group did not receive any treatment and were excluded from the safety population.) | 107 | 30
Completed | 81 | 27
Not Completed | 35 | 9
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 21 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 13 | 2

BASELINE CHARACTERISTICS:
Population: ITT Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With Radiesse | Untreated Control/Delayed Treatment With Radiesse | Total
Number analyzed (Participants) | 116 | 36 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (7.05) | 53.6 (8.08) | 53.6 (7.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 36 | 152
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 7 | 25
  Not Hispanic or Latino | 98 | 29 | 127
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 105 | 35 | 140
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders on Merz Aesthetic Scale (MAS) Décolleté Wrinkles - at Rest at Week 24
Description: The percentage of responders (responder rate) was defined as the percentage of subjects achieving greater than or equal to (>=) 1-point improvement on MAS décolleté wrinkles-at Rest from baseline to Week 24 as assessed by the blinded evaluator. Responder rate was assessed using MAS-at rest scale, where 0 = no wrinkles, 1 = mild wrinkles, 2 = moderate wrinkles, 3 = severe wrinkles, 4 = very severe wrinkles. Higher score indicated the worse outcome. This analysis was done using multiple imputation method to impute missing values.
Time Frame: Week 24
Population: ITT Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Treatment With Radiesse | Untreated Control/Delayed Treatment With Radiesse
Number analyzed (Participants) | 116 | 36
percentage of subjects | 71.2 [61.4 to 79.4] | 6.3 [1.5 to 22.9]
Statistical Analysis 1: Comparison: Treatment With Radiesse vs Untreated Control/Delayed Treatment With Radiesse; Test type: Superiority; Difference in response rates = 65.0, 95% CI 2-sided [45.6 to 74.4]

2. Secondary Outcome: Percentage of Responders on MAS Décolleté Wrinkles - Dynamic at Week 24
Description: The percentage of responders (responder rate) was defined as the percentage of subjects achieving >= 1-point improvement on MAS décolleté wrinkles-Dynamic from baseline to Week 24 as assessed by the blinded evaluator. Responder rate was assessed using MAS-Dynamic scale, where 0 = no wrinkles, 1 = mild wrinkles, 2 = moderate wrinkles, 3 = severe wrinkles, 4 = very severe wrinkles. Higher score indicated the worse outcome. This analysis was done using multiple imputation method to impute missing values.
Time Frame: Week 24
Population: ITT Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Treatment With Radiesse | Untreated Control/Delayed Treatment With Radiesse
Number analyzed (Participants) | 116 | 36
percentage of subjects | 65.8 [55.9 to 74.5] | 16.0 [6.8 to 33.1]

3. Secondary Outcome: Percentage of Subjects With Any Improvement on Investigator Global Aesthetic Improvement Scale (iGAIS) at Week 24
Description: Improvement is defined as a rating of +1 (Improved), +2 (Much improved) or +3 (Very much improved). Treating investigators used iGAIS, where - 3 = very much worse, - 2 = much worse, - 1 = worse, 0 = no change, + 1 = improved, + 2 = much improved, + 3 = very much improved. Higher score indicated aesthetic improvement.
Time Frame: Week 24
Population: ITT Analysis Set. Here "overall number of subjects analyzed" were the number of subjects with data available for analysis of this outcome measure at the given time point. This outcome measure was pre-specified and analyzed for subjects receiving Radiesse treatment only.
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment With Radiesse
Number analyzed (Participants) | 95
percentage of subjects | 92.6

4. Secondary Outcome: Percentage of Subjects With Any Improvement on Subject Global Aesthetic Improvement Scale (sGAIS) at Week 24
Description: Improvement is defined as a rating of +1 (Improved), +2 (Much improved) or +3 (Very much improved). Subjects used the sGAIS, where - 3 = very much worse, - 2 = much worse, - 1 = worse, 0 = no change, + 1 = improved, + 2 = much improved, + 3 = very much improved. Higher score indicated aesthetic improvement.
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment With Radiesse
Number analyzed (Participants) | 95
percentage of subjects | 87.4

5. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs) Related to Radiesse
Description: TEAEs are defined as AEs with onset on or after date of first administration of study treatment. Treatment related TEAEs are defined as any TEAEs related to diluted Radiesse treatment (that is, related to either injection procedure and/or device).
Time Frame: From initial treatment (Day 1 for Treatment group and Week 24 for Control/Delayed treatment group) up to end of the study (up to Week 84)
Population: SES included all subjects treated at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Radiesse | Untreated Control/Delayed Treatment With Radiesse
Number analyzed (Participants) | 107 | 30
Participants | 16 | 0

ADVERSE EVENTS:
Time Frame: From initial treatment (Day 1 for Treatment group and Week 24 for Control/Delayed treatment group) up to end of the study (up to Week 84)
Description: ITT Analysis set. The investigator reported AEs systematically at each visit.
Arm/Group | Treatment With Radiesse | Untreated Control/Delayed Treatment With Radiesse
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/36
Serious Adverse Events (participants affected / at risk) | 2/116 | 0/36
Other Adverse Events (participants affected / at risk) | 17/116 | 2/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Radiesse (N=116) | Untreated Control/Delayed Treatment With Radiesse (N=36)
Condition aggravated (General disorders) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Hip deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Radiesse (N=116) | Untreated Control/Delayed Treatment With Radiesse (N=36)
Visual acuity tests abnormal (Investigations) | 9 | 0
Injection site bruising (General disorders) | 7 | 0
COVID-19 (Infections and infestations) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT05163353/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT05163353/SAP_001.pdf